CLINICAL TRIAL: NCT06880133
Title: Evaluation and Improvement of Diagnostic Accuracy of Seismocardiography and Gyrocardiography for Non-Invasive Coronary Artery Disease Diagnosis in Comparison with Coronary Artery Calcium Computed Tomography, Coronary Computed Tomography Angiography, and Invasive Coronary Angiography
Brief Title: Expansion of SCG/GCG-Based CAD Sceering: Inclusion of Healthy Controls and CCTA Patients
Acronym: HF-CAD-CCTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Force Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UZ-Control-CCTA-1-16-02-388-19
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD))
Keywords: coronary artery disease; Seismocardiography; CardioClin
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SCG/GCG-Based CAD Screening with Healthy and CCTA Groups (Experimental): Participants in this arm will undergo seismocardiography (SCG) and gyrocardiography (GCG) testing to evaluate the diagnostic accuracy of these non-invasive methods in detecting coronary artery disease (CAD). SCG/GCG utilizes high-precision accelerometers and gyroscopes to measure cardiac-induced chest wall vibrations.
  This study will include patients scheduled for CAC-CT or CCTA at the Republic Specialized Scientific-Practical Medical Center of Cardiology (RSPCMCC). The primary goal is to determine whether SCG/GCG testing can predict CAD, particularly in patients with hypertension and mild or no CAD, by comparing SCG/GCG-derived data with standard imaging results.
  Measurements will be performed before CAC-CT and CCTA in both supine and upright sitting positions to assess the effect of posture on SCG/GCG signals.
  Interventions: Device: Seismocardiography (SCG) and Gyrocardiography (GCG) Screening

INTERVENTIONS:
Device: Seismocardiography (SCG) and Gyrocardiography (GCG) Screening — This intervention involves the use of SCG/GCG diagnostic testing, a radiation-free, non-invasive technique for assessing cardiac function. SCG/GCG utilizes high-precision accelerometers and gyroscopes to record and analyze cardiac-induced microvibrations on the chest.
  Participants will undergo SCG/GCG testing before their scheduled coronary artery calcium computed tomography (CAC-CT) or coronary computed tomography angiography (CCTA). The study aims to evaluate the diagnostic performance of SCG/GCG in identifying CAD, particularly in hypertensive patients and those with mild CAD.
  Data collected from SCG/GCG will be compared with CAC-CT and CCTA findings to determine its predictive value for CAD severity and coronary artery stenosis.

SUMMARY:
This study evaluates a new, non-invasive method for screening coronary artery disease (CAD) using seismocardiography (SCG) and gyrocardiography (GCG). These techniques measure chest vibrations caused by heart activity using highly sensitive sensors.

Participants include patients with known or suspected CAD, as well as healthy individuals and those undergoing coronary computed tomography angiography (CCTA). The goal is to determine whether SCG/GCG testing can accurately differentiate between individuals with significant and non-significant coronary artery stenosis.

SCG/GCG testing will be conducted before standard diagnostic procedures, including coronary artery calcium computed tomography (CAC-CT) and CCTA. The results will be analyzed to compare the performance of this novel method with existing imaging techniques.

This research aims to provide a non-invasive, cost-effective alternative for screening CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older.
* Electively scheduled for CAC-CT and have an indication for CCTA
* Suspected coronary artery disease (CAD) based on the presence of:
* At least two cardiovascular risk factors (e.g., hypertension, smoking, diabetes, dyslipidemia, obesity).
* CAD-related symptoms (e.g., chest pain, dyspnea on exertion).
* Suspected congenital coronary abnormalities.
* Ability to provide informed consent.

Exclusion Criteria:

* Severe cardiac arrhythmias that may interfere with SCG/GCG recordings.
* Decompensated heart failure or severe valvular heart disease.
* Other clinically significant concomitant diseases that may impact study participation.
* History of heart surgery (e.g., recent CABG, valve replacement) that alters chest wall dynamics.
* Contraindications for undergoing CAC-CT or CCTA (e.g., severe renal insufficiency preventing contrast use).
* Inability to remain still in supine or upright sitting positions for testing.
* Inability to provide informed consent due to cognitive or neurological conditions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Screening performance of SCG/GCG for Coronary Artery Disease (CAD) | Baseline
  The ability of Seismocardiography (SCG) and Gyrocardiography (GCG) testing to accurately detect coronary artery disease (CAD) compared to standard diagnostic methods (CCTA).

CONTACTS AND LOCATIONS:
Locations (1):
- Republic Specialized Scientific-Practical Medical Center of Cardiology (RSPCMCC), Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehkordi P, Bauer EP, Tavakolian K, Zakeri V, Blaber AP, Khosrow-Khavar F. Identifying Patients With Coronary Artery Disease Using Rest and Exercise Seismocardiography. Front Physiol. 2019 Sep 24;10:1211. doi: 10.3389/fphys.2019.01211. eCollection 2019. PMID 31607951
- [Background] Dehkordi P, Khosrow-Khavar F, Di Rienzo M, Inan OT, Schmidt SE, Blaber AP, Sorensen K, Struijk JJ, Zakeri V, Lombardi P, Shandhi MMH, Borairi M, Zanetti JM, Tavakolian K. Comparison of Different Methods for Estimating Cardiac Timings: A Comprehensive Multimodal Echocardiography Investigation. Front Physiol. 2019 Aug 22;10:1057. doi: 10.3389/fphys.2019.01057. eCollection 2019. PMID 31507437
- [Background] Dehkordi P, Tavakolian K, Tadi MJ, Zakeri V, Khosrow-Khavar F. Investigating the estimation of cardiac time intervals using gyrocardiography. Physiol Meas. 2020 Jun 10;41(5):055004. doi: 10.1088/1361-6579/ab87b2. PMID 32268315